CLINICAL TRIAL: NCT02380560
Title: Sonographic Assessment of Myometrial Thickness as a Predictor for the Latency Interval in Women With Preterm Premature Rupture of Membranes
Brief Title: Myometrial Thickness as a Predictor for the Latency Interval in PPROM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 129
Record Dates: First submitted 2015-02-26; First posted 2015-03-05 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Fetal Membranes, Premature Rupture
Keywords: myometrial thickness; Preterm premature rupture of membranes; Preterm Labour
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- pPROM: 50 women with preterm premature rupture of membranes with gestational age from 24 to 34 weeks assessed by ultrasound examination
  Interventions: Device: Ultrasonographic examination
- term non-labor control: 25 term non-labor control (T-CTR, n=25) with gestational age from 37 to 41 weeks assessed by ultrasound examination
  Interventions: Device: Ultrasonographic examination
- preterm non-labor control: 25 preterm non-labor control (P-CTR, n=25) with gestational age from 24 to 34 weeks assessed by ultrasound examination
  Interventions: Device: Ultrasonographic examination

INTERVENTIONS:
Device: Ultrasonographic examination — An abdominal ultrasound for: Estimation of gestational age, biophysical profile (BPP), Detection of any fetal gross anomalies, Assessment of fetal growth measurement of the Amniotic Fluid Index (AFI), Detection of any abnormal placental insertion and/or uterine structural abnormalities as septate or bicornuate uterus, measuring The myometrial thickness at 4 different sites:
  a) The lower uterine segment (LUS): 2cm above the reflection of the full urinary bladder (b)The anterior wall: 1cm above the maternal umbilicus. (c)Fundus: by placing the scan probe perpendicularly above the uterine fundus so that the entire curvature of the uterus is visualized.
  (d)The posterior wall: through using the maternal abdominal aortic pulsation as an anatomic marker.
  Other Names: obtetrics ultrasound

SUMMARY:
100 women divided into 3 groups:

* Group I: included 50 women with preterm premature rupture of membranes (PPROM, n=50) with gestational age from 24 to 34 weeks.
* Group II: included 25 term non-labor control (T-CTR, n=25) with gestational age from 37 to 41 weeks.
* Group III: included 25 preterm non-labor control (P-CTR, n=25) with gestational age from 24 to 34 weeks.The myometrial thickness at 4 different sites9:

  a) The lower uterine segment (LUS): 2cm above the reflection of the full urinary bladder (b)The anterior wall: 1cm above the maternal umbilicus. (c)Fundus: by placing the scan probe perpendicularly above the uterine fundus so that the entire curvature of the uterus was visualized.

  (d)The posterior wall: through using the maternal abdominal aortic pulsation as an anatomic marker.

At least 3 measurements were obtained at each site and averaged. The latency interval is determined in each of the 3 groups.

DETAILED DESCRIPTION:
The total number of pregnant women enrolled in the study was 100 women. These were divided into three groups:

* Group I: included 50 women with preterm premature rupture of membranes (PPROM, n=50) with gestational age from 24 to 34 weeks.
* Group II: included 25 term non-labor control (T-CTR, n=25) with gestational age from 37 to 41 weeks.
* Group III: included 25 preterm non-labor control (P-CTR, n=25) with gestational age from 24 to 34 weeks.Full History taking, including personal history for maternal age, obstetric history for number of previous pregnancies, history of previous PPROM. History of present pregnancy included gestational age, history of drug intake with special emphasis to women with PPROM giving history of gush of clear watery fluid from the vagina. Past history to exclude women with a contra- indication for conservative management in the study group.

Physical examinations: General examination for pulse, arterial blood pressure and temperature to exclude any signs of chorioamnionitis in the study group.

Abdominally, fundal level examinations for predicting the gestational age and/or IUGR or abnormalities of liquor. Monitoring of uterine contraction to pick up women who are not in labor in the study group.

P/V examination was not done for the three groups. While definite diagnosis of PPROM relied on sterile speculum examination showing a collection of fluid in the vagina. Some women needed direct observation of the cervix during a valsulva maneuver or with cough to show free flow of fluid from the cervical os.

Ultrasonographic examination: An abdominal ultrasound for: Estimation of gestational age, Assessment of fetal well being by biophysical profile (BPP), Detection of any fetal gross anomalies, Assessment of fetal growth to exclude IUGR, Sonographic estimation of fetal weight (SEFW), measurement of the Amniotic Fluid Index (AFI), Detection of any abnormal placental insertion and/or uterine structural abnormalities as septate or bicornuate uterus, measuring The myometrial thickness at 4 different sites9:

a) The lower uterine segment (LUS): 2cm above the reflection of the full urinary bladder (b)The anterior wall: 1cm above the maternal umbilicus. (c)Fundus: by placing the scan probe perpendicularly above the uterine fundus so that the entire curvature of the uterus was visualized.

(d)The posterior wall: through using the maternal abdominal aortic pulsation as an anatomic marker.

At least 3 measurements were obtained at each site and averaged. The latency interval is determined in each of the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy with a definite history of current PPROM for the study group

Exclusion Criteria:

* Suspected fetal growth restriction (IUGR),
* Any gross fetal anomalies,
* Abnormalities of placentation,
* Uterine structural abnormalities,
* Fetal jeopardy or intrauterine fetal death (IUFD).
* Women presenting with chorioamniointis with fever over 38 c abdominal tenderness, foul vaginal discharge and/or fetal tachycardia.
* Diabetics, immunocompromized and cardiac patients.
* Women with cervical cerclage.
* Women with drained liquor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The total number of pregnant women will be enrolled in the study is 100 women. These wwill be divided into three groups:
  * Group I: includes 50 women with preterm premature rupture of membranes (PPROM, n=50) with gestational age from 24 to 34 weeks.
  * Group II: includes 25 term non-labor control (T-CTR, n=25) with gestational age from 37 to 41 weeks.
  * Group III: includes 25 preterm non-labor control (P-CTR, n=25) with gestational age from 24 to 34 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
latency interval as determined sonographic myometrial thickness | weeks in gestation

SECONDARY OUTCOMES:
neonatal Apgar | 10 minutes after delivery
neonatal ICU admission | 24 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt